CLINICAL TRIAL: NCT06645834
Title: Smart MDI Randomized Controlled Trial in Subjects With Type 1 Diabetes (Smart MDI Study)
Brief Title: Smart MDI Study (CIP343)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP343
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Eligible subjects must successfully complete the run-in phase by demonstrating tolerance to sensor wear and compliance with study procedures prior to being randomized for the study phase, in which subjects will either be using the InPen™ with InPen™ App and Simplera™ system (Treatment Arm = T) or will continue under their MDI therapy with CGM (Control Arm = C) for another 6 months.
Masking Description: Not Applicable, No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Other): Subjects will start using the Smart MDI system consisting of the InPen™ System and Simplera™ System.
  Interventions: Device: Smart MDI System
- Control (No Intervention): None -Subjects will continue their own MDI therapy

INTERVENTIONS:
Device: Smart MDI System — The Smart MDI system consists of the InPen™ system and Simplera™ system.
  The InPen™ system includes a reusable smart bolus insulin pen injector with Bluetooth combined with the InPen™ app to help users take insulin doses.
  And InPen™ app which communicates with the InPen™ injector and compatible continuous glucose monitoring (CGM) devices to collect and display information on insulin delivered by the injector as well as current and past glucose values.
  The Simplera™ system consists of a disposable integrated sensor-transmitter platform (Simplera™ Sensor) and the Simplera™ app which receives data from the Simplera™ sensor via Bluetooth Low Energy (BLE) radio signal
  Arms: Treatment

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the Smart MDI system with InPen™ and Simplera™ in comparison with Multiple Daily Injection (MDI) therapy with intermittent scanning or real-time Continuous Glucose Monitoring (isCGM/CGM) over 6 months duration in people with type 1 diabetes to support the market access and therapy adoption of the Smart MDI system.

DETAILED DESCRIPTION:
This is a post-market, prospective, open-label, multi-center, randomized controlled trial in adult and pediatric subjects with type 1 diabetes.

The study consists of a run-in phase of 3 weeks and a study phase of 6 months.

The purpose of the run-in phase is to collect baseline HbA1c and CGM data while subjects are on their current therapy.

During the 6-month study phase, subjects will be randomized to continue with their current therapy or to start using the Smart MDI system.

Approximately 140 subjects with type 1 diabetes aged 2 years and older will be enrolled in the study at up to 20 investigational centers in Europe to achieve approximately 112 subjects randomized and completing the 6-month study phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 2 years or older at time of screening.
2. Subject is on MDI therapy (defined as ≥ 3 insulin injections per day and on a basal/bolus regimen) ≥ 6 months prior to screening.
3. Subject has a clinical diagnosis of type 1 diabetes for ≥ 12 months.
4. Subject is on MDI therapy with intermittent scanning or Continuous Glucose Monitoring (isCGM/CGM) ≥ 3 months prior to screening.
5. Subject has high compliance with sensor wear, per investigator assessment.
6. Subject has a Glycosylated hemoglobin (HbA1c) ≥ 8% (64 mmol/mol) as assessed locally at time of screening visit.
7. Subject is willing to take or switch to one of the InPen-compatible insulin types, NovoRapid™, Fiasp™, Humalog™ and Lyumjev™.
8. Subject or parent(s)/legal guardian(s) has a compatible mobile phone with Internet access.
9. Subject or parent(s)/legal guardian(s) is willing and able to provide written informed consent, comply with all study procedures and wear all study devices, as required during the study.

Exclusion Criteria:

1. Subject is using a Medtronic InPen™ for at least 3 months prior to screening.
2. Subject has untreated/unstable Addison's disease, growth hormone deficiency, hypopituitarism or definite gastroparesis, untreated coeliac disease, untreated thyroid disorder, or poorly controlled asthma, per investigator judgment.
3. Subject is planning to initiate or change to another glucose modifying therapy (for example pramlintide, DPP-4 inhibitor, GLP-1 agonists/mimetics, metformin or SGLT2 inhibitors).
4. Subject has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study chronically.
5. Subject has renal failure (stage 4 and above) defined by creatinine clearance of <30 ml/min, as assessed by Local Lab test ≤ 6 months before screening or performed at screening at Local Lab, as defined by the creatinine-based Cockcroft, CKD-EPI or MDRD equations.
6. Subject has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
7. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrollment into this study, as per investigator judgment.
8. Subject is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgment.
9. Subject has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
10. Subject is a woman of child-bearing potential who has a positive pregnancy test at screening or plans to become pregnant during the course of the study.
11. Subject is a woman who is breastfeeding.
12. Subject or parent(s)/legal guardian(s) is legally incompetent, illiterate or a vulnerable person.
13. Subject is a member of the research staff involved with executing the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 6-month study period
  The primary endpoint is the between-treatment (Smart MDI system arm vs MDI + isCGM or CGM arm) difference during the study phase in the percentage of time that the sensor glucose measurement is in the target range, 70 to 180 mg/dL (3.9-10.0 mmol/L). The endpoint will be assessed for non-inferiority with an absolute margin of 7.5% time in target range.

SECONDARY OUTCOMES:
Secondary Endpoint 1 | 6-month study period
  Mean HbA1c at the end of the 6-month study phase, non-inferiority test with an absolute margin of 0.4% HbA1c.
Secondary Endpoint 2 | 6-month study period
  % of Time spent in target range (70 to 180 mg/dL [3.9-10.0 mmol/L]) during the study phase, simple superiority test.
Secondary Endpoint 3 | 6-month study period
  Mean HbA1c at the end of the 6-month study phase, simple superiority test.

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (4):
  - Antwerp University Hospital, Antwerp
  - Hospital Universitaire Bruxelles Erasme, Brussels
  - UZ Leuven, Leuven
  - CHU Liege, Liège
- Czechia (2):
  - General University Hospital, Prague
  - IKEM, Prague
- France (4):
  - CHRU de Brest service diabetologie endocrinologie, Brest
  - Center for DIABeCare, Hospices Civils de Lyon, Lyon
  - CHU Nimes, Nîmes
  - Hospital Rangueil, Toulouse
- Germany (3):
  - Zentrum fur digitale Diabetologie Hamburg, Hamburg
  - Hannoversche Kinderheilanstalt, Hanover
  - MVZ Stoffwechselmedizin Leipzig, Leipzig
- Italy (2):
  - University of Bari Aldo Moro, Bari
  - ASST Spedali Civili Brescia, Brescia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Uddevalla Hospital, Uddevalla
  - Hogsbo Narsjukhus, Västra Frölunda

IPD SHARING:
Plan to Share IPD: No